CLINICAL TRIAL: NCT01490268
Title: Pharmacokinetic-pharmacodynamic Modeling of the Postoperative Pain Sensation During Patient-controlled Analgesia With Target-controlled Infusion of Hydromorphone, Taking Into Account the Interaction With Intraoperatively Administered Sufentanil for Elective Cardiac Surgery
Brief Title: Pain Therapy After Elective Cardiac Surgery
Acronym: PKPDHM-001
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PKPDHM-001; 2011-003648-31 (EudraCT Number)
Record Dates: First submitted 2011-11-28; First posted 2011-12-12 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Pain
Keywords: Pharmacokinetic-pharmacodynamic modeling; Patient-controlled analgesia; Target-controlled infusion; Hydromorphone; Sufentanil; after thoracotomy; cardiac surgery
MeSH Terms: conditions — Pain | interventions — Sufentanil; Hydromorphone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sufentanil Group 1 (Active Comparator): Sufentanil Low Titration
  Interventions: Drug: Sufentanil, Hydromorphone
- Sufentanil Group 2 (Active Comparator): Sufentanil High Titration
  Interventions: Drug: Sufentanil, Hydromorphone

INTERVENTIONS:
Drug: Sufentanil, Hydromorphone — Intraoperatively: Target controlled infusion with 0.4 ng/ml Sufentanil, Postoperatively: Patient-controlled analgesia with target-controlled infusion of Hydromorphone
  Arms: Sufentanil Group 1
Drug: Sufentanil, Hydromorphone — Intraoperatively: Target controlled infusion with 0.8 ng/ml Sufentanil, Postoperatively: Patient-controlled analgesia with target-controlled infusion of Hydromorphone
  Arms: Sufentanil Group 2

SUMMARY:
The purpose of this study is to determine generation of a target controlled infusion model for the patient controlled analgesia with the strong analgesic, hydromorphone, after planned open heart surgery, during which the strong analgesic, sufentanil, was used.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent,
* Ability to understand the nature of patient-controlled analgesia and other study-specific procedures,
* Elective cardiac surgery with thoracotomy and subsequent stay in the intensive care unit

Exclusion Criteria:

* Use of MAO inhibitors in the last 14 days,
* Chronic alcoholism or drug addiction in medical history,
* Severe obstructive or restrictive pulmonal disorders in medical history,
* Severe hepatic and renal disorders in medical history,
* Hypothyroidism, pancreatitis in medical history,
* ASA IV,
* Pregnant or nursing females

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-11; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of sufentanil and hydromorphone | 48 hours
  28 blood samples are taken during the study period of 48 hours postoperatively for characterizing the pharmacokinetics
Numerical Rating Scale for Clinical Pain | 8 hours
  11 assessments of patient's pain sensation using Numerical Rating Scale for Clinical Pain during patient-controlled analgesia with target-controlled infusion of hydromorphone 8 hours after extubation for characterizing the analgesic effect

SECONDARY OUTCOMES:
Total amount of hydromorphone | 8 hours
  Cumulative dose of hydromorphone for patient-controlled analgesia with target-controlled infusion of hydromorphone for characterizing the analgesic requirement
Modified Observer's Assessment of Alertness/Sedation (MOAA/S) Scale | 8 hours
  11 assessments of the Modified Observer's Assessment of Alertness/Sedation (MOAA/S) Scale during patient-controlled analgesia with target-controlled infusion of hydromorphone 8 hours after extubation for characterizing the sedation level

CONTACTS AND LOCATIONS:
Overall Officials: Christian Jeleazcov, MD, Principal Investigator — Department of Anesthesiology, University Hospital Erlangen, Germany
Locations (1):
- Department of Anesthesiology, University Hospital, Erlangen, Germany

REFERENCES:
- [Background] Jeleazcov C, Saari TI, Ihmsen H, Mell J, Frohlich K, Krajinovic L, Fechner J, Schuttler J. Population pharmacokinetic modeling of hydromorphone in cardiac surgery patients during postoperative pain therapy. Anesthesiology. 2014 Feb;120(2):378-91. doi: 10.1097/ALN.0b013e3182a76d05. PMID 23958818
- [Background] Saari TI, Ihmsen H, Mell J, Frohlich K, Fechner J, Schuttler J, Jeleazcov C. Influence of intensive care treatment on the protein binding of sufentanil and hydromorphone during pain therapy in postoperative cardiac surgery patients. Br J Anaesth. 2014 Oct;113(4):677-87. doi: 10.1093/bja/aeu160. Epub 2014 Jul 6. PMID 25001621
- [Background] Saari TI, Fechner J, Ihmsen H, Schuttler J, Jeleazcov C. Analysis of total and unbound hydromorphone in human plasma by ultrafiltration and LC-MS/MS: application to clinical trial in patients undergoing open heart surgery. J Pharm Biomed Anal. 2012 Dec;71:63-70. doi: 10.1016/j.jpba.2012.07.025. Epub 2012 Jul 31. PMID 22884788
- [Background] Saari TI, Fechner J, Ihmsen H, Schuttler J, Jeleazcov C. Determination of total and unbound sufentanil in human plasma by ultrafiltration and LC-MS/MS: application to clinical pharmacokinetic study. J Pharm Biomed Anal. 2012 Jul;66:306-13. doi: 10.1016/j.jpba.2012.03.050. Epub 2012 Apr 3. PMID 22522038